CLINICAL TRIAL: NCT01331655
Title: A Multicenter, Open-label, 3-arm, Active-controlled, Parallel-group, 1-year Study to Investigate the Efficacy and Safety of a Flexible Regimen of the Combined Oral Contraceptive, With and Without 0.451 mg Levomefolate Calcium (BAY98-7071 and BAY86-5300, Respectively) Versus the Standard 24 + 4 Regimen With Levomefolate (BAY98-7071 + BAY86-7660) and to Assess Compliance With a Device (CADDY) in Healthy Women Who Desire Contraception
Brief Title: Clinical Study of a Conventional and Flexible Extended Oral Contraceptive of EE/DRSP With or Without Metafolin in Latin America
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14700
Record Dates: First submitted 2011-04-07; First posted 2011-04-08 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Contraception
MeSH Terms: interventions — 5-methyltetrahydrofolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: EE20/DRSP (BAY86-5300)
- Arm 2 (Experimental)
  Interventions: Drug: EE20/DRSP/L-5-MTHF (BAY98-7071)
- Arm 3 (Active Comparator)
  Interventions: Drug: EE20/DRSP/L-5-MTHF (BAY98-7071) + L-5-MTHF (BAY86-7660)

INTERVENTIONS:
Drug: EE20/DRSP (BAY86-5300) — Day 1-120: 0.02 mg EE as ß-CDC / 3 mg DRSP (1 tablet/day); up to 120-day treatment period followed by a 4-day tablet-free interval
  Arms: Arm 1
Drug: EE20/DRSP/L-5-MTHF (BAY98-7071) — Day 1-120: 0.02 mg EE as ß-CDC / 3 mg DRSP / 0.451 mg levomefolate calcium (1 tablet/day) up to 120-day treatment period followed by a 4-day tablet-free interval
  Arms: Arm 2
Drug: EE20/DRSP/L-5-MTHF (BAY98-7071) + L-5-MTHF (BAY86-7660) — Day 1-24: 0.02 mg EE as ß-CDC / 3 mg DRSP / 0.451 mg levomefolate calcium per tablet (1 tablet/day) Day 25-28: tablets with 0.451 mg levomefolate calcium (1 tablet/day)
  Arms: Arm 3

SUMMARY:
The objective of this three-arm study is to evaluate the effect of a flexible extended regimen of an EE+DRSP containing OC on bleeding pattern and to investigate the compliance with daily pill intake when the investigational product is provided in a blister package or a compliance aiding dispenser with a pill reminder function. The third treatment arm will be a reference comparator arm of a standard 24+4 regimen of the identical hormone combination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers between 18 and 35 years of age (smokers up to 30 years, inclusive) who request contraceptive protection

Exclusion Criteria:

* Pregnancy or lactation (less than 3 months since delivery, abortion, or lactation before start of treatment)
* Body mass index (BMI) >/= 30.0 kg/m2
* Presence or a history of venous or arterial thrombotic/thromboembolic events
* Repeated measurements of systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg
* Presence or history of liver tumors (benign or malignant), severe hepatic disease, jaundice and/or pruritus related to cholestasis, cholestatic jaundice associated with pregnancy or previous combined oral contraceptive (COC) use
* Uncontrolled diabetes mellitus and/or diabetes mellitus with vascular involvement
* Severe dyslipoproteinemia
* Malignant or premalignant disease
* Uncontrolled thyroid disorder
* Chronic inflammatory bowel disease

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Number of bleeding days | Approximately 1 year

SECONDARY OUTCOMES:
Difference in the number of missed tablets between Arms A and B | Approximately 1 year
Bleeding pattern and cycle control parameters | Approximately 1 year
Number of cycles per subject | Approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer